CLINICAL TRIAL: NCT03886961
Title: The Effect of the Reflux Band™ Upper Esophageal Sphincter (UES) Assist Device on Reflux for Lung Transplant Recipients
Acronym: Reflux Band
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Somna Therapeutics, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB201900469 -A
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Lung Transplant; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lung Transplant Patients (Experimental): For the first four weeks, lung transplant patients will not wear the Reflux Band. Use of the Reflux Band will subsequently commence in the next four weeks.
  Interventions: Device: Reflux Band

INTERVENTIONS:
Device: Reflux Band — The Reflux Band is to be worn when sleeping by lung transplant patients for 4 weeks starting 8 weeks after transplant.
  Other Names: Reflux Band™ Upper Esophageal Sphincter (UES) Assist Device

SUMMARY:
A prospective, open label, study designed to assess the affect of the Reflux Band® UES Assist Device (Reflux Band) on reflux in patients that have undergone lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable lung transplant patients(single lung, double lung, or re-transplant) as defined by stable FEV1 over the prior two visits
* 13 Abnormal pH impedence or esophagram or documented gastric reflux at pre-transplant evaluation
* Patient must be willing and able to provide informed consent
* Understands the clinical study requirements and is able to comply with follow-up schedule

Exclusion Criteria:

* Currently being treated with another investigational medical device and/or drug
* Currently receiving treatment for sleep apnea with continuous positive airway pressure (CPAP)
* Previous head or neck surgery / radiation
* Carotid artery disease, thyroid disease, or history of cerebral vascular disease
* Nasopharyngeal cancer
* Suspected esophageal cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-17 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in pepsin levels | Baseline; Week 4; Week 8
  The presence of reflux will be assessed by measuring levels of pepsin in bronchoalveolar lavage fluid.
Change in amylase levels | Baseline; Week 4; Week 8
  The presence of reflux will be assessed by measuring levels of amylase in bronchoalveolar lavage fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Amaris, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No